CLINICAL TRIAL: NCT05776472
Title: A Single Arm, Long-term, Multicentre Observational Study to Evaluate Effectiveness of Pegcetacoplan Under Real World Conditions in Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Brief Title: A Real World Effectiveness Study of Pegcetacoplan in Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Acronym: COMPLETE
Status: Recruiting | Type: Observational
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: Sobi.PEGCET-304
Record Dates: First submitted 2023-02-20; First posted 2023-03-20 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — pegcetacoplan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Pegcetacoplan — Pegcetacoplan will be prescribed according to the label in patients with PNH.
  Other Names: Aspaveli, Empaveli

SUMMARY:
This is a 36-month, long-term, multicenter, observational study designed to describe the real world effectiveness of pegcetacoplan in patients with PNH. Patients meeting the eligibility criteria will be enrolled in the study and followed prospectively for approximately 36 months. Patient data will be collected from start of pegcetacoplan treatment to end of follow-up. Retrospective data on pegcetacoplan will be captured from the time of pegcetacoplan treatment initiation. Pegcetacoplan treatment data will be collected for a minimum of approximately 36 months and up to a maximum of approximately 72 months, including retrospective period depending on when the patient started pegcetacoplan treatment. After pegcetacoplan treatment discontinuation, patients will remain in the study for 8 weeks to capture any AEs. The scope of the study is to collect both retrospective and prospective data. Baseline is defined as start of pegcetacoplan treatment. The main part of the study will be prospective,collecting data on effectiveness, safety (all AEs), patient- and clinician-reported outcomes and health care resource use.

DETAILED DESCRIPTION:
As pegcetacoplan is a new product on the market, with a new mechanism of action, there is an urgent need to provide data to treaters, payers and the PNH community on the real-world usage and effectiveness of pegcetacoplan. This study aims to fill part of that knowledge gap and to add to the knowledge base regarding the use of pegcetacoplan in routine medical practice. Another important rationale for this study is to provide information on RBC transfusions and health care resource utilization pre and post pegcetacoplan treatment initiation.

The study plans to include approximately 200 patients at 70 sites in Europe, Middle East, Canada and Australia. Additional countries may be added in the study if necessary. Patients meeting the eligibility criteria will be enrolled in the study and followed prospectively for approximately 36 months. Patient data will be collected from start of pegcetacoplan treatment to end of follow-up. Retrospective data on pegcetacoplan will be captured from the time of pegcetacoplan treatment initiation. Pegcetacoplan treatment data will be collected for a minimum of approximately 36 months and up to a maximum of approximately 72 months, including retrospective period depending on when the patient started pegcetacoplan treatment. After pegcetacoplan treatment discontinuation, patients will remain in the study for 8 weeks to capture any AEs. Patients will come to their routine visits and the available data from each visit will be collected.

The scope of the study is to collect both retrospective and prospective data. The main part of the study will be prospective, collecting data on effectiveness, safety, patient- and clinician-reported outcomes and health care resource use. The study will also collect retrospective data before pegcetacoplan treatment start, which will consist of information on PNH treatment, blood transfusions and healthcare resource use. Data will be collected for up to 12 months prior to pegcetacoplan treatment start. As patients may have been treated with pegcetacoplan for up to 12 months prior to enrollment, retrospective data may be collected for up to 24 months. This means that the total data collection period including both the retrospective and the prospective part is up to 48 (+/- 3) months.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age with a documented PNH diagnosis.
* Patient started routine treatment with pegcetacoplan for PNH up to 12 months before enrollment or prescribed pegcetacoplan at enrollment. Decision to initiate treatment shall be made by the treating physician and independently from the decision to include the patient in the study.
* Patient is willing and able to provide written informed consent to participate in the study in a manner approved by the Institutional Review Board/Independent Ethics Committee and local regulations.

Exclusion Criteria:

* Enrollment in a concurrent clinical interventional study, or intake of an Investigational Medicinal Product (IMP), within three months prior to the start of the current pegcetacoplan treatment.
* Initiated current treatment with pegcetacoplan in an interventional study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) with PNH, who started routine treatment with pegcetacoplan up to 12 months prior to enrollmentor at enrollment
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2029-08-15 (Estimated)

PRIMARY OUTCOMES:
Change in observed hemoglobin level from initiation of treatment with pegcetacoplan to 6 months | 6 months
  Hemoglobin level in g/dL.

SECONDARY OUTCOMES:
Change of LDH values from initiation of pegcetacoplan treatment to 6 months | 6 months
  Lactate Dehydrogenase (LDH) in U/L
Change in Absolute Reticulocyte Count (ARC) from initiation of pegcetacoplan treatment to 6 months | 6 months
  Absolute Reticulocyte Count (ARC) in 10^9/L
Change in indirect/ total bilirubin from initiation of pegcetacoplan treatment to 6 months | 6 months
  Indirect/ total bilirubin in umol/L
Change in Haptoglobin from initiation of pegcetacoplan treatment to 6 months | 6 months
  Haptoglobin in mg/dL
Change in Ferritin from initiation of pegcetacoplan treatment to 6 months | 6 months
  Ferritin in ug/L
Hemoglobin at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 6 months
  Hemoglobin in g/dL
Hemoglobin at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 12 months
  Hemoglobin in g/dL
Hemoglobin at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 18 months
  Hemoglobin in g/dL
Hemoglobin at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 24 months
  Hemoglobin in g/dL
Hemoglobin at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 30 months
  Hemoglobin in g/dL
Hemoglobin at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 36 months
  Hemoglobin in g/dL
Lactate Dehydrogenase at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 6 months
  Lactate Dehydrogenase (LDH) in U/L
Lactate Dehydrogenase at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 12 months
  Lactate Dehydrogenase (LDH) in U/L
Lactate Dehydrogenase at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 18 months
  Lactate Dehydrogenase (LDH) in U/L
Lactate Dehydrogenase at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 24 months
  Lactate Dehydrogenase (LDH) in U/L
Lactate Dehydrogenase at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 30 months
  Lactate Dehydrogenase (LDH) in U/L
Lactate Dehydrogenase at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 36 months
  Lactate Dehydrogenase (LDH) in U/L
Absolute Reticulocyte Count at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 6 months
  Absolute Reticulocyte Count (ARC) in 10^9/L
Absolute Reticulocyte Count at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 12 months
  Absolute Reticulocyte Count (ARC) in 10^9/L
Absolute Reticulocyte Count at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 18 months
  Absolute Reticulocyte Count (ARC) in 10^9/L
Absolute Reticulocyte Count at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 24 months
  Absolute Reticulocyte Count (ARC) in 10^9/L
Absolute Reticulocyte Count at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 30 months
  Absolute Reticulocyte Count (ARC) in 10^9/L
Absolute Reticulocyte Count at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 36 months
  Absolute Reticulocyte Count (ARC) in 10^9/L
Indirect/ total bilirubin at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 6 months
  Indirect/ total bilirubin in umol/L
Indirect/ total bilirubin at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 12 months
  Indirect/ total bilirubin in umol/L
Indirect/ total bilirubin at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 18 months
  Indirect/ total bilirubin in umol/L
Indirect/ total bilirubin at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 24 months
  Indirect/ total bilirubin in umol/L
Indirect/ total bilirubin at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 30 months
  Indirect/ total bilirubin in umol/L
Indirect/ total bilirubin at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 36 months
  Indirect/ total bilirubin in umol/L
Haptoglobin at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 6 months
  Haptoglobin in µmol/L
Haptoglobin at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 12 months
  Haptoglobin in µmol/L
Haptoglobin at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 18 months
  Haptoglobin in µmol/L
Haptoglobin at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 24 months
  Haptoglobin in µmol/L
Haptoglobin at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 30 months
  Haptoglobin in µmol/L
Haptoglobin at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 36 months
  Haptoglobin in mg/dL
Ferritin at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 6 months
  Ferritin in ug/L
Ferritin at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 12 months
  Ferritin in ug/L
Ferritin at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 18 months
  Ferritin in ug/L
Ferritin at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 24 months
  Ferritin in ug/L
Ferritin at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 30 months
  Ferritin in ug/L
Ferritin at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 36 months
  Ferritin in ug/L
Hemoglobin ≥ 12 g/dL at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 6 months
  Hemoglobin in g/dL
Hemoglobin ≥ 12 g/dL at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 12 months
  Hemoglobin in g/dL
Hemoglobin ≥ 12 g/dL at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 18 months
  Hemoglobin in g/dL
Hemoglobin ≥ 12 g/dL at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 24 months
  Hemoglobin in g/dL
Hemoglobin ≥ 12 g/dL at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 30 months
  Hemoglobin in g/dL
Hemoglobin ≥ 12 g/dL at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 36 months
  Hemoglobin in g/dL
Increase in hemoglobin levels of ≥ 2 g/dL at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 6 months
  Hemoglobin in g/dL
Increase in hemoglobin levels of ≥ 2 g/dL at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 12 months
  Hemoglobin in g/dL
Increase in hemoglobin levels of ≥ 2 g/dL at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 18 months
  Hemoglobin in g/dL
Increase in hemoglobin levels of ≥ 2 g/dL at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 24 months
  Hemoglobin in g/dL
Increase in hemoglobin levels of ≥ 2 g/dL at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 30 months
  Hemoglobin in g/dL
Increase in hemoglobin levels of ≥ 2 g/dL at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 36 months
  Hemoglobin in g/dL
Hemolytic event requiring additional intervention at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 6 months
  Yes/No
Hemolytic event requiring additional intervention at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 12 months
  Yes/No
Hemolytic event requiring additional intervention at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 18 months
  Yes/No
Hemolytic event requiring additional intervention at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 24 months
  Yes/No
Hemolytic event requiring additional intervention at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 30 months
  Yes/No
Hemolytic event requiring additional intervention at initiation of pegcetacoplan treatment and each 6 months until end of follow-up | 36 months
  Yes/No
Annualized number of red blood cell (RBC) transfusions during pegcetacoplan treatment until end of follow-up compared to the 12 month period before pegcetacoplan treatment | 12 months
  Total number of RBC transfusions
Annualized number of red blood cell (RBC) units during pegcetacoplan treatment until end of follow-up compared to the 12 month period before pegcetacoplan treatment | 12 months
  Total number of RBC units
Fatigue at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 6 months
  Patient reported outcome scale scores for the Functional assessment of chronic illness therapy (FACIT) - Fatigue. It is a 13-item scale and each item is scored on a 5-point Likert Scale ranging from "0-Not at all" to "4-Very much". The FACIT-fatigue score is obtained by summing all item scores. The score range from 0 to 52, higher score indicating less fatigue and lower score indicating more fatigue.
Fatigue at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 12 months
  Patient reported outcome scale scores for the Functional assessment of chronic illness therapy (FACIT) - Fatigue. It is a 13-item scale and each item is scored on a 5-point Likert Scale ranging from "0-Not at all" to "4-Very much". The FACIT-fatigue score is obtained by summing all item scores. The score range from 0 to 52, higher score indicating less fatigue and lower score indicating more fatigue.
Fatigue at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 18 months
  Patient reported outcome scale scores for the Functional assessment of chronic illness therapy (FACIT) - Fatigue. It is a 13-item scale and each item is scored on a 5-point Likert Scale ranging from "0-Not at all" to "4-Very much". The FACIT-fatigue score is obtained by summing all item scores. The score range from 0 to 52, higher score indicating less fatigue and lower score indicating more fatigue.
Fatigue at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 24 months
  Patient reported outcome scale scores for the Functional assessment of chronic illness therapy (FACIT) - Fatigue. It is a 13-item scale and each item is scored on a 5-point Likert Scale ranging from "0-Not at all" to "4-Very much". The FACIT-fatigue score is obtained by summing all item scores. The score range from 0 to 52, higher score indicating less fatigue and lower score indicating more fatigue.
Fatigue at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 30 months
  Patient reported outcome scale scores for the Functional assessment of chronic illness therapy (FACIT) - Fatigue. It is a 13-item scale and each item is scored on a 5-point Likert Scale ranging from "0-Not at all" to "4-Very much". The FACIT-fatigue score is obtained by summing all item scores. The score range from 0 to 52, higher score indicating less fatigue and lower score indicating more fatigue.
Fatigue at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 36 months
  Patient reported outcome scale scores for the Functional assessment of chronic illness therapy (FACIT) - Fatigue. It is a 13-item scale and each item is scored on a 5-point Likert Scale ranging from "0-Not at all" to "4-Very much". The FACIT-fatigue score is obtained by summing all item scores. The score range from 0 to 52, higher score indicating less fatigue and lower score indicating more fatigue.
Health care resource use: Annualized number of hospitalizations and emergency room visits during pegcetacoplan treatment until end of follow-up compared to the 12-month period before pegcetacoplan treatment. | 12 months
  Number of hospitalizations and emergency room visits
Patient treatment satisfaction every 6 months until end of follow-up | 6 months
  Patient treatment satisfaction (1-5 point scale), 5=highly satisfied, 1= highly dissatisfied
Patient treatment satisfaction every 6 months until end of follow-up | 12 months
  Patient treatment satisfaction (1-5 point scale), 5=highly satisfied, 1= highly dissatisfied
Patient treatment satisfaction every 6 months until end of follow-up | 18 months
  Patient treatment satisfaction (1-5 point scale), 5=highly satisfied, 1= highly dissatisfied
Patient treatment satisfaction every 6 months until end of follow-up | 24 months
  Patient treatment satisfaction (1-5 point scale), 5=highly satisfied, 1= highly dissatisfied
Patient treatment satisfaction every 6 months until end of follow-up | 30 months
  Patient treatment satisfaction (1-5 point scale), 5=highly satisfied, 1= highly dissatisfied
Patient treatment satisfaction every 6 months until end of follow-up | 36 months
  Patient treatment satisfaction (1-5 point scale), 5=highly satisfied, 1= highly dissatisfied
Physician treatment satisfaction every 6 months until end of follow-up | 6 months
  Physician treatment satisfaction (1-5 point scale), 5=highly satisfied, 1= highly dissatisfied
Physician treatment satisfaction every 6 months until end of follow-up | 12 months
  Physician treatment satisfaction (1-5 point scale), 5=highly satisfied, 1= highly dissatisfied
Physician treatment satisfaction every 6 months until end of follow-up | 18 months
  Physician treatment satisfaction (1-5 point scale), 5=highly satisfied, 1= highly dissatisfied
Physician treatment satisfaction every 6 months until end of follow-up | 24 months
  Physician treatment satisfaction (1-5 point scale), 5=highly satisfied, 1= highly dissatisfied
Physician treatment satisfaction every 6 months until end of follow-up | 30 months
  Physician treatment satisfaction (1-5 point scale), 5=highly satisfied, 1= highly dissatisfied
Physician treatment satisfaction every 6 months until end of follow-up | 36 months
  Physician treatment satisfaction (1-5 point scale), 5=highly satisfied, 1= highly dissatisfied
Adverse events (AE), including serious adverse events (SAE) | 24 hours
  Adverse events (AE) and serious adverse events (SAE) are to be reported on the AE page of the eCRF as specified in the eCRF data entry guidelines.
Alanine transaminase (ALT) at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 6 months
  Alanine transaminase (ALT) in U/L
Alanine transaminase (ALT) at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 12 months
  Alanine transaminase (ALT) in U/L
Alanine transaminase (ALT) at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 18 months
  Alanine transaminase (ALT) in U/L
Alanine transaminase (ALT) at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 24 months
  Alanine transaminase (ALT) in U/L
Alanine transaminase (ALT) at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 30 months
  Alanine transaminase (ALT) in U/L
Alanine transaminase (ALT) at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 36 months
  Alanine transaminase (ALT) in U/L
Aspartate aminotransferase (AST) at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 6 months
  Aspartate aminotransferase (AST) in U/L
Aspartate aminotransferase (AST) at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 12 months
  Aspartate aminotransferase (AST) in U/L
Aspartate aminotransferase (AST) at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 18 months
  Aspartate aminotransferase (AST) in U/L
Aspartate aminotransferase (AST) at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 24 months
  Aspartate aminotransferase (AST) in U/L
Aspartate aminotransferase (AST) at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 30 months
  Aspartate aminotransferase (AST) in U/L
Aspartate aminotransferase (AST) at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 36 months
  Aspartate aminotransferase (AST) in U/L
Alkaline Phosphatase at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 6 months
  Alkaline Phosphatase in µkat/L
Alkaline Phosphatase at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 12 months
  Alkaline Phosphatase in µkat/L
Alkaline Phosphatase at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 18 months
  Alkaline Phosphatase in µkat/L
Alkaline Phosphatase at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 24 months
  Alkaline Phosphatase in µkat/L
Alkaline Phosphatase at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 30 months
  Alkaline Phosphatase in µkat/L
Alkaline Phosphatase at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 36 months
  Alkaline Phosphatase in µkat/L
Bilirubin at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 6 months
  Indirect/ total bilirubin in umol/L
Bilirubin at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 12 months
  Indirect/ total bilirubin in umol/L
Bilirubin at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 18 months
  Indirect/ total bilirubin in umol/L
Bilirubin at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 24 months
  Indirect/ total bilirubin in umol/L
Bilirubin at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 30 months
  Indirect/ total bilirubin in umol/L
Bilirubin at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 36 months
  Indirect/ total bilirubin in umol/L
Creatinine at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 6 months
  Creatinine in mg/dL
Creatinine at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 12 months
  Creatinine in mg/dL
Creatinine at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 18 months
  Creatinine in mg/dL
Creatinine at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 24 months
  Creatinine in mg/dL
Creatinine at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 30 months
  Creatinine in mg/dL
Creatinine at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 36 months
  Creatinine in mg/dL
estimated glomerular filtration rate (eGFR) at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 6 months
  estimated glomerular filtration rate (eGFR) in mL/min/1.73 m²
estimated glomerular filtration rate (eGFR) at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 12 months
  estimated glomerular filtration rate (eGFR) in mL/min/1.73 m²
estimated glomerular filtration rate (eGFR) at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 18 months
  estimated glomerular filtration rate (eGFR) in mL/min/1.73 m²
estimated glomerular filtration rate (eGFR) at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 24 months
  estimated glomerular filtration rate (eGFR) in mL/min/1.73 m²
estimated glomerular filtration rate (eGFR) at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 30 months
  estimated glomerular filtration rate (eGFR) in mL/min/1.73 m²
estimated glomerular filtration rate (eGFR) at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 36 months
  estimated glomerular filtration rate (eGFR) in mL/min/1.73 m²
Urea at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 6 months
  Urea in mg/dL
Urea at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 12 months
  Urea in mg/dL
Urea at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 18 months
  Urea in mg/dL
Urea at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 24 months
  Urea in mg/dL
Urea at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 30 months
  Urea in mg/dL
Urea at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 36 months
  Urea in mg/dL
Potassium at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 6 months
  Potassium in mmol/L
Potassium at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 12 months
  Potassium in mmol/L
Potassium at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 18 months
  Potassium in mmol/L
Potassium at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 24 months
  Potassium in mmol/L
Potassium at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 30 months
  Potassium in mmol/L
Potassium at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 36 months
  Potassium in mmol/L
Sodium at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 6 months
  Sodium in mmol/L
Sodium at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 12 months
  Sodium in mmol/L
Sodium at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 18 months
  Sodium in mmol/L
Sodium at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 24 months
  Sodium in mmol/L
Sodium at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 30 months
  Sodium in mmol/L
Sodium at initiation of treatment with pegcetacoplan and every 6 months until end of follow-up | 36 months
  Sodium in mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Study Physician +46 08-697-20 00, medical.info@sobi.com, Study Director — Swedish Orphan Biovitrum
Locations (75):
- Australia (3):
  - Liverpool Hospital, Liverpool, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
- Belgium (4):
  - AZ Sint-Jan, Bruges
  - CHU Brugmann-Site Horta, Brussels
  - Centre Hospitalier Universitaire de Liege, Liège
  - AZ Turnhout - Campus Sint-Elisabeth, Turnhout
- Canada (2):
  - University Health Network, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont d/b/a CIUSSS de l'Est-de-l'Île-de-Montréal, Montreal, Quebec
- Czechia (2):
  - Fakultni nemocnice Brno, Brno
  - Ustav hematologie a krevni transfuze, Prague
- Helsingin yliopistollinen keskussairaala, Helsinki, Finland
- France (10):
  - CHU Nice - Hôpital de l'Archet 1, Nice, Alpes Maritimes
  - CHU de Bordeaux - Hôpital Haut-Lévêque, Pessac, Gironde
  - Hopital Foch, Suresnes, Hauts De Seine
  - CHU de Grenoble - Hôpital Albert Michallon, Grenoble, Isere
  - CHU de Nantes - Hotel Dieu, Nantes, Loire Atlantique
  - CHU de Nancy - Hôpital de Brabois Adultes, Vandœuvre-lès-Nancy, Meurthe Et Moselle
  - Hopital Claude Huriez - CHRU Lille, Lille, Nord
  - Hôpital Saint-Louis, La Defense, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Rhone
  - CHU Poitiers, Poitiers
- Germany (9):
  - Alb-Fils-Kliniken GmbH, Goettigen, Baden-Wurttemberg
  - Studienzentrum Aschaffenburg, Aschaffenburg, Bavaria
  - Universitaetsklinikum Frankfurt Goethe-Universitaet, Frankfurt am Main, Hesse
  - Universitaetsklinikum Giessen und Marburg GmbH Standort Giessen, Giessen, Hesse
  - Dres Ballo und Dr. Böck, Offenbach, Hesse
  - Universitaetsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitaetsklinikum Leipzig AoeR, Leipzig, Saxony
  - Praxis Fenchel Saalfeld, Saalfeld, Thuringia
  - MV Zentrum für Onkologie und Hämatologie, Cologne
- Greece (5):
  - Evangelismos Hospital, Athens
  - University General Hospital "Attikon", Athens
  - University General Hospital of Larissa, Larissa
  - G Papanikolaou General Hospital, Thessaloniki
  - General Hospital of Thessaloniki "IPPOKRATEIO", Thessaloniki
- Hungary (3):
  - DPC - Orszagos Hematologiai es Infektologiai Intezet, Budapest
  - Semmelweis Egyetem, Budapest
  - Semmelweis University, Budapest
- Italy (12):
  - Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari, Bari
  - Ospedale San Bassiano, Bassano del Grappa
  - Irccs Aou Di Bologna- Pol. Di S.Orsola, Bologna
  - Ospedale Oncologico Armando Businco, Cagliari
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale San Raffaele, Milan
  - Ospedale Maggiore della Carità, Novara
  - Grande Ospedale Metropolitano - Presidio Morelli, Reggio Calabria
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Università di Roma La Sapienza, Rome
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino, Torino
- Poland (7):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Szpital Uniwersytecki nr 2 im. dr J. Biziela w Bydgoszczy, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - SPZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - WWCOiT in Lodz, Oddział Hematologii i Transplantologii, Lodz
  - Uniwersytecki Szpital Kliniczny nr 1 w Lublinie, Lublin
  - Warszawski Uniwersytet Medyczny, Warsaw
- Saudi Arabia (4):
  - Prince Faisal Bin Bandar Cancer Center, Buraidah
  - King Faisal Specialist Hospital & Research Center, Jeddah
  - King Faisal Specialist Hospital and Research Center - Madinah, Riyadh
  - King Faisal Specialist Hospital and Research Center - Riyadh, Riyadh
- Spain (12):
  - ICO Badalona - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital de Cruces, Barakaldo
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Hospital Universitario Virgen de la Nieves, El Palmar
  - Hospital Universitario de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
  - Hospital Lucus Augusti, Lugo
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Central de Asturias, Oviedo
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No